CLINICAL TRIAL: NCT05558046
Title: Predictive Value of Granulosa Cell DNA Damage in the Success of Assisted Reproductive Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Erman Çiftçi, MD, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Other Study IDs: 07/2022
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: DNA Damage; Granulosa Cells
Keywords: Ovarian Reserve; Flow Cytometry; Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Granulosa cells will be isolated by using hyaluronidase. A single cell suspension will be obtained by filtering through 70 micron pores. The cells will be centrifuged remove the supernatants and the cells will be suspended in phosphate buffered saline (PBS). CD45+ cells which will be suspended in PBS will be labeled with Pacific Blue fluorochrome-conjugated anti-CD45 antibody. The cells will be fixed with 1% paraformaldehyde, the fixative solution will be removed and permeabilized with PBS containing 0.1% Triton X-100 and 1% bovine serum albumin (BSA) block solution. Fixation and permeabilization stages, both processes will be carried out at 4°C. Permeabilized cells will be suspended in PBS containing 1% BSA, with Alexa Fluor 700 fluorochrome-conjugated Histone H2A.X and Alexa Fluor 488 fluorochrome-conjugated Gamma H2A.X antibodies at 4°C. The cells will be read using the DxFLEX flow cell meter system. The protein levels of Histone H2A.X and its phosphorylated form will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Ovarian Reserve: Patients diagnosed as low ovarian reserve were recruited to the study who have Antimüllerian Hormone level of 1 ng/ml or lower. Patients with low ovarian reserve were diagnosed after normal standard infertility evaluation according to the guideline of The Practice Committee of the American Society for Reproductive Medicine which consist of the assesment of spermiogram, ovulation, hysterosalpingogram and if indicated ovarian reserve tests and laparoscopy. Male infertility is an exclusion.
- Unexplained Infertile (Control group): Patients diagnosed as unexplained infertility (UI) were recruited to the study who have Antimüllerian Hormone level of 1.5 ng/ml or higher as a control group. UI was diagnosed after normal standard infertility evaluation according to the guideline of The Practice Committee of the American Society for Reproductive Medicine which consist of the assesment of spermiogram, ovulation, hysterosalpingogram and if indicated ovarian reserve tests and laparoscopy.

SUMMARY:
Deoxyribonucleic acid (DNA) damage of granulosa cells obtained during oocyte retrieval will be evaluated by flow cytometry with detection of Histone H2A.X and Phosphorylated Gamma H2A.X protein levels in patients with low ovarian reserve and unexplained infertile patients as a control group undergoing intracytoplasmic sperm injection (ICSI) treatment. Fertilization, embryo quality, transfer rate, implantation, clinical pregnancy will be recorded as well as demographic data. DNA damage of granulosa cells will be compared between two groups. The effect of DNA damage of granulosa cells on fertilization, quality of oocyte and embryo, implantation, and clinical pregnancy will be also evaluated.

DETAILED DESCRIPTION:
Granulosa cells surrounding the oocytes will be mechanically obtained during the oocyte pick-up procedure in women undergoing intracytoplasmic sperm injection (ICSI) treatment due to unexplained infertility and low ovarian reserve. Deoxyribonucleic acid (DNA) damage in these cells will be evaluated by flow cytometry. Fertilization rates, embryo quality by grading, and transfer rates will also be assessed. Implantation and clinical pregnancy rates will be recorded as well as demographic data such as age, body-mass index, smoking, alcohol use, employment, coexisting chronic disease, infertility duration, etiology of infertility, treatment protocol. Implantation will be evaluated by determination of serum human chorionic gonadotropin (hCG) at day 15 following an embryo transfer. Clinical pregnancy will be diagnosed upon presence of gestational sac on ultrasound examination. DNA damage of granulosa cells will be compared between low ovarian reserve group and control group. The effect of DNA damage of granulosa cells on fertilization, quality of oocyte and embryo, implantation, and clinical pregnancy will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* For patients who are undergoing in Vitro Fertilization (IVF) treatment with Low ovarian reserve, Antimullerian Hormone level must be lower than 1 ng/mL
* For patients who are undergoing in Vitro Fertilization (IVF) treatment with Unexplained infetility, Antimullerian Hormone level must be greater than 1,5 ng/mL

Exclusion Criteria:

* Chronic systemic disease (rheumatoid arthritis, hypertension, diabetes..)
* Endocrinopathy (Thyroid, prolactin... abnormalities)
* Chemotherapy or radiotherapy history
* Endometriosis
* Policystic ovary syndrome
* Male infetility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients ages between 18 years to 35 years
Study Population: Low ovarian reserve group will be included as Antimullerian hormone level results as lower than 1 ng/ml without any other infertility evidence.The control group received IVF for Unexplained infertile (UI) group UI was diagnosed after normal standard infertility evaluation according to the guideline of The Practice Committee of the American Society for Reproductive Medicine which consist of the assesment of spermiogram, ovulation, hysterosalpingogram and if indicated ovarian reserve tests and laparoscopy as well as Antimullerian hormone level results as greater than 1,5 ng/ml. If the results of all this tests were normal, patients were accepted as UI.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Determining the correlation of ovarian reserve and age factor with DNA Damage markers in granulosa cells. | 1 day
  Demographic data will be noted for each patient at the day of oocyte retrieval, and DNA damage markers will be shown by flowcytometry at the same day.

SECONDARY OUTCOMES:
Fertilization defined as the presence of two pronuclei under light microscope one day after intracytoplasmic sperm injection procedure | 1 day after ICSI procedure
  Presence of two pronuclei under light microscope
Implantation defined as positive serum human chorionic gonadotropin levels 12 days after embryo transfer | 12 days after embryo transfer
  Positive human chorionic gonadotropin levels
Clinical pregnancy will be defined as the presence of gestational sac in transvaginal ultrasonographic examination 5 weeks after embryo transfer | 5 weeks
  Presence of a gestational sac in transvaginal ultrasonographic examination